CLINICAL TRIAL: NCT00002394
Title: A Four-Week, Open-Label, Non-Randomized, Multicenter, Dose-Finding, Pilot Study to Evaluate the Safety and Efficacy of Two Daily Doses of Lamisil (1500 Mg and 2000 Mg), Administered for a Maximum of 4 Weeks in HIV-Positive Subjects With Oral Mucosal Candidiasis Not Having Responded to a Minimum of 200 Mg Fluconazole Monotherapy
Brief Title: Safety and Effectiveness of Giving Lamisil to HIV-Positive Subjects With Thrush Who Have Not Responded to Fluconazole Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novartis (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 282A; SFS 257-E-00
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-12

CONDITIONS: Candidiasis, Oral; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Dose-Response Relationship, Drug; Fluconazole; Antifungal Agents; Candidiasis, Oral; Drug Administration Schedule; terbinafine
MeSH Terms: conditions — Candidiasis, Oral; HIV Infections; AIDS-Related Opportunistic Infections | interventions — Terbinafine

INTERVENTIONS:
Drug: Terbinafine hydrochloride

SUMMARY:
The purpose of this study is to see if it is safe and effective to give Lamisil to HIV-positive patients with thrush (a fungal infection) that has not responded to fluconazole.

DETAILED DESCRIPTION:
This is an open-label, dose-escalating study with up to 2 sequential cohorts. The first 15 patients receive Lamisil for 2 weeks. After 2 weeks, patients considered clinically cured (i.e., absence of removable, white plaques) are removed from treatment; patients not considered clinically cured receive an additional 2 weeks of treatment. At the end of 4 weeks, treatment is discontinued, regardless of clinical cure outcome. If less than 80% of patients are clinically cured after the 4 weeks of treatment, a second cohort of 15 patients receive Lamisil on the same treatment regimen as first cohort (i.e., initial 2-week treatment period, with an additional 2 weeks of treatment for those patients who are not considered clinically cured after 2 weeks of treatment).

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are at least 18 years old.
* Have thrush that has not responded to at least 10 days of fluconazole treatment.
* Are HIV-positive.
* Are expected to live at least 4 weeks.
* Are able to take oral medication.

Exclusion Criteria

You will not be eligible for this study if you:

* Have liver or kidney disease.
* Have received certain medications.
* Have a history of serious diarrhea or digestive problems.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Therafirst Med Ctr, Fort Lauderdale, Florida
  - Associates in Research, Fort Myers, Florida
  - Clireco Inc, Tamarac, Florida
  - Infectious Diseases Research Inc, Tampa, Florida
  - Northwestern Univ / Division of Infectious Disease, Chicago, Illinois
  - Saint Michaels Med Ctr / Infectious Disease Resch Dpt, Newark, New Jersey
  - St Vincents Hosp / Clinical Research Program, New York, New York
  - Univ of Texas Med Branch, Galveston, Texas
  - Hampton Roads Med Specialists, Hampton, Virginia